CLINICAL TRIAL: NCT03538444
Title: A Double-Blind, Randomized, Controlled Trial, Utilizing Accelerated Repetitive Transcranial Magnetic Stimulation (rTMS) as a Tool to Decrease Pain and Craving in Hospitalized Patients With Opiate Use Disorder
Brief Title: Repetitive Transcranial Magnetic Stimulation for Opiate Use Disorder
Acronym: ArTMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment stopped due to COVID19 and PI made an institution switch.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00077611
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Opiate Dependence; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: 40 individuals (20 per group) will be randomly assigned to either active or sham rTMS.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither participants nor investigators will know whether the participant is assigned to the active or sham condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active rTMS (Experimental): Participants will receive 18 sessions of active repetitive Transcranial Magnetic Stimulation over a period of three days. TMS consists of 3000 pulses of 10Hz stimulation applied to the left DLPFC using the beam F3 method
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Placebo Comparator): Participants will receive 18 sessions of sham rTMS over a period of three days.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation technique which is currently FDA-approved as a treatment for major depressive disorder
  Other Names: Active rTMS
  Arms: Active rTMS
Device: Sham rTMS — Participants will undergo procedures that mimic rTMS, but that are inactive.
  Arms: Sham rTMS

SUMMARY:
This double-blind, randomized, controlled trials will investigate the effect of accelerated, repeated transcranial magnetic stimulation on opiate craving and perceived pain .

DETAILED DESCRIPTION:
Prescription opiate use disorder (OUD) is common in the United States, with high morbidity and mortality. Despite the availability of opiate replacement therapies, many individuals continue to abuse opiates and relapse rates remain high. Uncontrolled pain and opiate craving are both commonly reported by OUD individuals attempting abstinence, and likely contribute to relapse. As such, development of novel treatment strategies targeting pain and craving would have important clinical implications.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation technique which is currently FDA-approved as a treatment for major depressive disorder. TMS is actively being pursued as a treatment for chronic pain disorders as well as for substance use disorders. In chronic pain patients, there is promising data suggesting that treatment with excitatory rTMS to the dorsolateral pre-frontal cortex (DLPFC) can have an anti-pain effect. A single session of excitatory DLPFC rTMS can decrease the perception of laboratory induced pain, decrease the amount of self administered morphine following open gastric bypass surgery and decrease the affective and sensory components of pain following laparoscopic gastric-bypass surgery. While the effects of a single session last for only approximately 1 hour, repeated sessions appear to have an additive and more durable effect, and following 15 sessions, the subjective experience of provoked pain has been shown to decrease by as much as 37%. In addition to the literature in laboratory induced pain, there is also preliminary data suggesting that rTMS may be an effective treatment for chronic pain disorders. In substance use disordered populations, the use of rTMS has garnered significant attention as an innovative tool to decrease craving [see reviews:. Several single session rTMS studies have demonstrated that applying excitatory rTMS to the DLPFC can decrease cue-induced craving in nicotine, cocaine, and alcohol use disordered populations. As expected, single session studies have only found small temporary reductions in craving; however, these promising data have led to preliminary clinical trials using multiple sessions of rTMS in alcohol, nicotine and cocaine use disorders. The largest such clinical trial (n=130 smokers) demonstrated that 13 sessions of DLPFC rTMS resulted in six month tobacco abstinence rates of 33% .

To date there has been limited work examining the effect of rTMS on craving or pain in individuals with OUD. Drawing from the published literature suggesting that excitatory rTMS applied to the DLPFC can reduce both pain and craving, our group completed a preliminary sham-controlled crossover study in prescription OUD patients with chronic pain. Our data suggest that a single session of excitatory DLPFC rTMS acutely decreased opiate cue induced craving and thermal pain sensitivity in this group. The promising results from our single session trial parallel the single session results found in nicotine and cocaine use disordered populations which subsequently translated into positive multiple session clinical trials. As such, it follows that a trial utilizing multiple sessions of rTMS in OUD patients may yield positive results.

40 participants (20/group) admitted to an inpatient community treatment facility for opiate detoxification will be given 18 sessions of either active or sham rTMS applied to the DLPFC, in an accelerated fashion over three days (6-sessions each day).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
2. Participants must meet DSM-5 criteria for moderate or severe OUD. While individuals may also meet criteria for use disorders of other substances (with the exception of alcohol or benzodiazepines), they must identify prescription opiates as their primary substance of abuse.
3. Participants must be admitted to the inpatient unit for opiate detoxification.
4. Participants must consent to random assignment.

Exclusion Criteria:

1. Participants who are pregnant will be excluded.
2. Participants with a history of/or current psychotic disorder will be excluded.
3. Participants with a history of dementia or other cognitive impairment will be excluded.
4. Participants with active suicidal ideation, or a suicide attempt within the past 90 days will be excluded.
5. Participants with contraindications to receiving rTMS (including a history of seizures, or any implanted metal above the neck) will be excluded.
6. Those with unstable general medical conditions will be excluded.
7. Those who are currently using naltrexone, or tramadol, will be excluded.
8. Those with alcohol or benzodiazepine use disorders will be excluded due to increased risk of seizure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active rTMS | Sham rTMS
Started | 4 | 3
Completed | 3 | 3
Not Completed | 1 | 0
Not completed — opioid withdrawal | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS | Sham rTMS | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (2) | 36 (13.1) | 31.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7
Composite Provoked Opioid Craving 0-30 likert scale (sum of 0-10 each for want, resist, crave) [Mean (Standard Deviation); unit: units on a scale, higher -> more craving] | 11 (6.9) | 23.7 (8.5) | 19.1 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: Composite Opioid Craving (Want, Resist, Crave)
Description: Change in cue-induced craving ratings on 10 point Likert Scales. 0=Not at all; 10=Extremely How much do you WANT TO USE _(opiate of choice)_ right now? HOW HARD would it be for you TO RESIST USING_(opiate of choice)_ right now if it was offered to you? How much do you currently crave opiates? (scores on each of those questions are summed to be between 0 and 30 with 30 being the highest (and indicating the most craving).
Time Frame: Baseline and three days: Pre-assessment (day 1-prior to the first delivered rTMS treatment) compared to post assessment (AM of day4 the morning following the final of three days of rTMS)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 3 | 3
units on a scale | 0.7 (1.2) | 16.7 (12.7)

ADVERSE EVENTS:
Time Frame: 1-month
Description: As per clinicaltrials.gov definitions
Arm/Group | Active rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/4 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS (N=4) | Sham rTMS (N=3)
headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT03538444/Prot_SAP_002.pdf